CLINICAL TRIAL: NCT01690416
Title: Conventional vs Ultrasound Guided Arteria Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Marlene A Hansen, Stud.med, Stud.med, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: sloth2; Overlæge Dr. Med Edgar Schnohr (Other Grant/Funding Number: Overlæge Dr. Med Edgar Schnohr)
Record Dates: First submitted 2012-09-13; First posted 2012-09-21 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Disorder of Cardiac Function

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound DNTP (Active Comparator): the catheter will be placed using ultrasound and DNTT and Lidocaine as local anesthesia, by the same fellow as the one who performs the puncture with the traditional method
  Interventions: Procedure: Traditional palpation technique; Procedure: Ultrasound DNTP
- Traditional palpation technique (Active Comparator): arteria cannulation by traditional palpation technique, using preprocedural lidocaine for anesthetic and palpation method by a fellow
  Interventions: Procedure: Traditional palpation technique; Procedure: Ultrasound DNTP

INTERVENTIONS:
Procedure: Traditional palpation technique
Procedure: Ultrasound DNTP

SUMMARY:
The aim of the project is to compare two methods for arterial cannulation. The traditional method with ultrasound guided cannulation. The investigators goal is to improve this procedure to reduce pain and complications.

DETAILED DESCRIPTION:
The practice of placing vascular catheters is used many times every day at almost every hospital. It is a safe procedure which generally does not imply problems. Though the procedural optimum aren't reached. The procedure still fails some times and induce complications. When the catheter is placed using the traditional method the pulse is palpated by the operator's fingers. This is only to be done near the hand wrist. In this position the catheter steadiness is fragile but because the pulse can't be sensed more proximal the operator is forced to choose this position. This it though a problem that can be solved by non invasive visualization technology. Ultrasound-guidance for central vascular access is already well-established. However, in recent years ultrasound-guidance for peripheral vascular access has gained popularity too. The evidence of multiple studies demonstrates increased success rate and reduced complication rate with ultrasound compared to blind landmark technique for vascular catheter placement.

In recent years there have been both procedural technique and technology improvements in the field of ultrasound. This has led to the improvement of procedural catheterisation techniques that now can be done by novices with higher attempt success rate than traditional method. One technique that is gaining success is the short-axis-out-of-plane technique (SAX-OOP) with dynamic-needle-tip-tracking (DNTT).Using the ultrasound machine the needle can be placed in a more proximal direction on the forearm and the investigators believe that by the help of the exposed procedure on the monitor many complications can be reduced.

It has been shown that inexperienced trainees lear the technique SAX-OOP and DNTT very quickly.

First investigators hypothesize that the number of attempts, the number of withdrawals, the time spend and the number of utilized catheters will be decreased using ultrasound vs. the traditional method. Secondly investigators hypothesize that the pain induced by the conventional method inclusive preoperational lidocaine injection will be the same or more intense than using DNTT with local anesthesia. Thirdly investigators claim that the best anatomical place to put the catheter isn't always corresponding with the spot chosen by palpation, which increase the number of failures. Fourthly investigators hypothesize that the use of ultrasound will increase the operator's subjective feeling of having accomplished a successful procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-90 years
* Fulfill the criteria of an operation
* Routine need of an arterial needle

Exclusion Criteria:

* Lack of patient consent
* Ultrasound identified plaques in the radial artery or ultrasound verified compromised flow in either the radial or ulnar artery.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Attempts | 1 hour
  The number of attempts (skin punctures) per catheterization
Withdrawals | 1 hour
  The number of withdrawals of the guide-needle per catheterization
Time consume | minutes
  The time spend for the catheterization procedure
Catheters | 1 hour
  The number of utilized catheters

SECONDARY OUTCOMES:
pain | momentan
  The pain induced by the conventional method inclusive preoperational lidocaine injection will be the same or more intense than using DNTT with local anesthesia measured on a VAS-score.
Ease of method for the operator | momentan
  The use of ultrasound will increase the operator's subjective feeling of having accomplished a successful procedure on a Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Aa Hansen, stud.med, Principal Investigator — Anæstesiologisk-Intensiv afd I
Locations (1):
- Aarhus Universitets Hospital, Aarhus, Jylland, Denmark